CLINICAL TRIAL: NCT02463760
Title: Predicting Rupture of Abdominal Aortic Aneurysm (AAA) by Anatomic and Hemodynamic Markers From In-vivo and In-vitro Imaging
Brief Title: Predicting Rupture of AAA by Anatomic and Hemodynamic Markers
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 150023
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical imaging

SUMMARY:
The purpose of the study is to investigate imaging findings, which can help us to predict factors contributing to abdominal aortic aneurysm growth and rupture.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 80 years old receiving medical care at University of Minnesota Medical Center who have a normal aorta CTA within the previous year
* Or patients with known AAA with growth rate of 0-0.2 cm/year
* Or patients with known AAA with growth rate of greater than 0.5 cm/year.

Exclusion Criteria:

* Subjects with ferromagnetic implants
* Penile implant
* Hip replacement
* History of shrapnel or shot gun injury
* Body mass index ≥ 30
* Cardiac pacemakers
* Severe claustrophobia
* Large tattoos on the torso

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary and specialty care clinics and emergency room visits.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Imaging findings correlating with abdominal aortic aneurysm growth and rupture | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosenberg, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided